CLINICAL TRIAL: NCT03112460
Title: Cardiopulmonary Resuscitation Training Program Based on Quality Control in Gottsegen György Hungarian Institute of Cardiology
Brief Title: Cardiopulmonary Resuscitation Training Program Based on Quality Control
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hungarian Institute of Cardiology (Other Government)
Responsible Party: Principal Investigator, ANDREKA PETER, Head of Department of Cardiology, Hungarian Institute of Cardiology
Other Study IDs: CPRTPBQC
Record Dates: First submitted 2017-03-17; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Cardiopulmonary Resuscitation
MeSH Terms: interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- all patients: all of patients who went through basic and advanced cardiopulmonary resuscitations would be analyzed
  Interventions: Device: cardiopulmonary resuscitation with Zoll R Series defibrillator and defibrillator pads with a real-time CPR feedback option and CodeReview case analysis software

INTERVENTIONS:
Device: cardiopulmonary resuscitation with Zoll R Series defibrillator and defibrillator pads with a real-time CPR feedback option and CodeReview case analysis software — cardiopulmonary resuscitation with Zoll R Series defibrillator and defibrillator pads with a real-time CPR feedback option and CodeReview case analysis software

SUMMARY:
In a prospective, non-randomized study, all of the basic and advanced cardiopulmonary resuscitations would be analyzed. All resuscitation are planned to be performed by the above mentioned devices according to the recent protocols. The continuous audio-visual feedback and all the data obtained during the resuscitation are intended to develop a better CPR training program in the future.

The downloading of data is planned to occur on the same day of CPR to a data card. After approximately one week all the participant medical persons would receive a detailed case analysis. Elimination of the typical errors is targeted.

Monitored quality indicators

Follow-up of CPR protocol:

elapsed time between turning on device and first chest compression elapsed time between turning on device and first delivered shock elapsed time between turning on device and first delivered shock in case of shockable rhythm compliance with 2 minutes long CPR period recognition of rhythm, recognition of adequate therapy, follow-up of the protocol concerning DC-shock recording the exact moment of the following procedures (with the use of Code Marker button on the defibrillator device) endotracheal intubation drug therapy obtaining intravenous access oxygen therapy

Quality of chest compressions:

depth frequency release compression fraction

Discontinuance of chest compression - cause anf time interval (Code Marker) endotracheal intubation ventilation rhythm analysis and defibrillation obtaining intravenous access

Other data (obtaining with manual recording):

cause of sudden cardiac death initial rhythm exact time of sudden death eyewitness records data of the patient monitoring system (only optional) description of place participant of CPR first detection medical documentation

DETAILED DESCRIPTION:
Sudden cardiac death remains the leading cause of morbidity and mortality and has public health importance. In recent decades, the pathophysiology became better known, however despite the development of medical devices and therapies, significant improvement in outcome was not observed, survival of patients remained low REF1-4.

The resuscitation protocols are based on universal algorithms REF5-6, are valid for all health care practitioners regardless of qualifications, skills. This reanimation paradigm focuses on the basic skills (chest compression, respiration) REF7-8. On the basis of investigations, the most important factors would be: continuous, high-quality chest compressions with the possibly of shortest interruptions REF9, however, the performance of this practice has significant difficulties to meet the expectations REF10.

Without relevant data, the meaningful assessment, follow-up and analysis of resuscitation are difficult, so a substantive case-based training is not feasible.

A reanimation training program on the basis of continuous audio-visual feedback, data and case report would be needed to improve the poor outcome.

A study proved that audio-visual cardiopulmonary resuscitation (CPR) feedback, case analysis and scenario-based training can improve significantly the parameters of basic life support (BLS) and can increase the odds of a better neurological survival status after sudden cardiac arrest outside a hospital - adjusted odds ratio (AOR) 2.7 REF11.

Another study REF12 demonstrated that this method in a hospital environment can improve CPR quality indicators. The so-called Advanced Resuscitation the framework program has also achieved a significant leap from the hospital survival (AOR 2.2, good neurological status AOR 3.0) with similar methods and technology REF13. These results show that an increase in the survival can be achieved with the improvement of resuscitation method and training.

Advanced life support (ALS) service in the Gottsegen György Hungarian Institute of Cardiology is provided by the medical staff of the Cardiology Intensive Care Unit (emergency medical team - EMT).

Our aim is to evolve a continuous quality improvement program with the usage of ZOLL R Series defibrillator device and defibrillator pads with a real-time CPR feedback option and CodeReview case analysis software, and to provide further execution of the program thereafter.

In a prospective, non-randomized study, all of the basic and advanced cardiopulmonary resuscitations would be analyzed. All resuscitation are planned to be performed by the above mentioned devices according to the recent protocols. The continuous audio-visual feedback and all the data obtained during the resuscitation are intended to develop a better CPR training program in the future.

The downloading of data is planned to occur on the same day of CPR to a data card. After approximately one week all the participant medical persons would receive a detailed case analysis. Elimination of the typical errors is targeted.

Monitored quality indicators

Follow-up of CPR protocol:

elapsed time between turning on device and first chest compression elapsed time between turning on device and first delivered shock elapsed time between turning on device and first delivered shock in case of shockable rhythm compliance with 2 minutes long CPR period recognition of rhythm, recognition of adequate therapy, follow-up of the protocol concernig DC-shock recording the exact moment of the following procedures (with the use of Code Marker button on the defibrillatior device) endotracheal intubation drug therapy obtaining intravenous access oxygen therapy

Quality of chest compressions:

depth frequency release compression fraction

Discontinuance of chest compression - cause anf time interval (Code Marker) endotracheal intubation ventilation rhythm analysis and defibrillation obtaining intravenous access

Other data (obtaining with manual recording):

cause of sudden cardiac death initial rhythm exact time of sudden death eyewitness records data of the patient monitoring system (only optional) description of place participant of CPR first detection medical documentation

Participant of the study:

Péter ANDRÉKA Prof. MD, Head of Department, Principal Investigator of study Gábor UZONYI MD, Head of Intensive Care Unit Krisztina SZÜTS MD András CSEPREGI MD Attila KOVÁCS MD Péter TAKÁCS MD András BECK MD Csaba SÁRI MD, Coordinator of study Adrienn MANDZÁK MD Judit POLANECZKY Anna NAGYNÉ LŐKE

ELIGIBILITY:
inclusion criteria: all-cause circulatory arrest exclusion criteria: "do not resuscitate" code, age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who went through basic and advanced cardiopulmonary resusciations would be analyzed
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-07-31 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Follow-up of CPR protocol | period of cardiopulmonary resuscitation (up to 2 hours)
  elapsed time between turning on device and first chest compression elapsed time between turning on device and first delivered shock elapsed time between turning on device and first delivered shock in case of shockable rythm compliance with 2 minutes long CPR period recognition of rythm, recognition of adequate therapy, follow-up of the protocol concernig DC-shock recording the exact moment of the following procedures (with the use of Code Marker button on the defibrillatior device)
Quality of chest compressions | period of cardiopulmonary resuscitation (up to 2 hours)
  depth frequency release compression fraction
Discontinuance of chest compression - cause anf time interval (Code Marker) | period of cardiopulmonary resuscitation (up to 2 hours)
  endotracheal intubation ventilation rythm analysis and defibrillation obtaning intravenous access

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dans PE, Nevin KL, Seidman CE, McArthur JC, Kariya ST. Inhospital CPR 25 years later: why has survival decreased? South Med J. 1985 Oct;78(10):1174-8. PMID 4049035
- [Background] Sasson C, Rogers MA, Dahl J, Kellermann AL. Predictors of survival from out-of-hospital cardiac arrest: a systematic review and meta-analysis. Circ Cardiovasc Qual Outcomes. 2010 Jan;3(1):63-81. doi: 10.1161/CIRCOUTCOMES.109.889576. Epub 2009 Nov 10. PMID 20123673
- [Background] Nichol G, Thomas E, Callaway CW, Hedges J, Powell JL, Aufderheide TP, Rea T, Lowe R, Brown T, Dreyer J, Davis D, Idris A, Stiell I; Resuscitation Outcomes Consortium Investigators. Regional variation in out-of-hospital cardiac arrest incidence and outcome. JAMA. 2008 Sep 24;300(12):1423-31. doi: 10.1001/jama.300.12.1423. PMID 18812533
- [Background] Peberdy MA, Kaye W, Ornato JP, Larkin GL, Nadkarni V, Mancini ME, Berg RA, Nichol G, Lane-Trultt T. Cardiopulmonary resuscitation of adults in the hospital: a report of 14720 cardiac arrests from the National Registry of Cardiopulmonary Resuscitation. Resuscitation. 2003 Sep;58(3):297-308. doi: 10.1016/s0300-9572(03)00215-6. PMID 12969608
- [Background] Monsieurs KG, Nolan JP, Bossaert LL, Greif R, Maconochie IK, Nikolaou NI, Perkins GD, Soar J, Truhlar A, Wyllie J, Zideman DA; ERC Guidelines 2015 Writing Group. European Resuscitation Council Guidelines for Resuscitation 2015: Section 1. Executive summary. Resuscitation. 2015 Oct;95:1-80. doi: 10.1016/j.resuscitation.2015.07.038. Epub 2015 Oct 15. No abstract available. PMID 26477410
- [Background] Perkins GD, Jacobs IG, Nadkarni VM, Berg RA, Bhanji F, Biarent D, Bossaert LL, Brett SJ, Chamberlain D, de Caen AR, Deakin CD, Finn JC, Grasner JT, Hazinski MF, Iwami T, Koster RW, Lim SH, Ma MH, McNally BF, Morley PT, Morrison LJ, Monsieurs KG, Montgomery W, Nichol G, Okada K, Ong ME, Travers AH, Nolan JP; Utstein Collaborators. Cardiac Arrest and Cardiopulmonary Resuscitation Outcome Reports: Update of the Utstein Resuscitation Registry Templates for Out-of-Hospital Cardiac Arrest: A Statement for Healthcare Professionals From a Task Force of the International Liaison Committee on Resuscitation (American Heart Association, European Resuscitation Council, Australian and New Zealand Council on Resuscitation, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa, Resuscitation Council of Asia); and the American Heart Association Emergency Cardiovascular Care Committee and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. Resuscitation. 2015 Nov;96:328-40. doi: 10.1016/j.resuscitation.2014.11.002. Epub 2014 Nov 11. PMID 25438254
- [Background] Neumar RW, Otto CW, Link MS, Kronick SL, Shuster M, Callaway CW, Kudenchuk PJ, Ornato JP, McNally B, Silvers SM, Passman RS, White RD, Hess EP, Tang W, Davis D, Sinz E, Morrison LJ. Part 8: adult advanced cardiovascular life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S729-67. doi: 10.1161/CIRCULATIONAHA.110.970988. PMID 20956224
- [Background] Sayre MR, Koster RW, Botha M, Cave DM, Cudnik MT, Handley AJ, Hatanaka T, Hazinski MF, Jacobs I, Monsieurs K, Morley PT, Nolan JP, Travers AH; Adult Basic Life Support Chapter Collaborators. Part 5: Adult basic life support: 2010 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2010 Oct 19;122(16 Suppl 2):S298-324. doi: 10.1161/CIRCULATIONAHA.110.970996. No abstract available. PMID 20956253
- [Background] Abella BS, Sandbo N, Vassilatos P, Alvarado JP, O'Hearn N, Wigder HN, Hoffman P, Tynus K, Vanden Hoek TL, Becker LB. Chest compression rates during cardiopulmonary resuscitation are suboptimal: a prospective study during in-hospital cardiac arrest. Circulation. 2005 Feb 1;111(4):428-34. doi: 10.1161/01.CIR.0000153811.84257.59. PMID 15687130
- [Background] Bobrow BJ, Vadeboncoeur TF, Stolz U, Silver AE, Tobin JM, Crawford SA, Mason TK, Schirmer J, Smith GA, Spaite DW. The influence of scenario-based training and real-time audiovisual feedback on out-of-hospital cardiopulmonary resuscitation quality and survival from out-of-hospital cardiac arrest. Ann Emerg Med. 2013 Jul;62(1):47-56.e1. doi: 10.1016/j.annemergmed.2012.12.020. Epub 2013 Mar 7. PMID 23465553
- [Background] Crowe C, Bobrow BJ, Vadeboncoeur TF, Dameff C, Stolz U, Silver A, Roosa J, Page R, LoVecchio F, Spaite DW. Measuring and improving cardiopulmonary resuscitation quality inside the emergency department. Resuscitation. 2015 Aug;93:8-13. doi: 10.1016/j.resuscitation.2015.04.031. Epub 2015 May 8. PMID 25963706
- [Background] Davis DP, Graham PG, Husa RD, Lawrence B, Minokadeh A, Altieri K, Sell RE. A performance improvement-based resuscitation programme reduces arrest incidence and increases survival from in-hospital cardiac arrest. Resuscitation. 2015 Jul;92:63-9. doi: 10.1016/j.resuscitation.2015.04.008. Epub 2015 Apr 20. PMID 25906942